CLINICAL TRIAL: NCT04504227
Title: Effect of Thickened Feeds on Swallow Physiology in Children With Dysphagia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Daniel Duncan, Assistant Professor of Pediatrics, Boston Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: IRB-P00036103; K23DK127251 (NIH)
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-02

CONDITIONS: Dysphagia; Aspiration; Brief Resolved Unexplained Event (BRUE); Apparent Life Threatening Event (ALTE)
MeSH Terms: conditions — Deglutition Disorders; Brief, Resolved, Unexplained Event

STUDY DESIGN:
Intervention Model Description: 4-test consistency, randomized, crossover, single-blinded swallow physiology study comparing effects of different liquid viscosities on swallow coordination in infants and children
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Thin liquid swallows (Placebo Comparator): Thin liquid swallows of formula or breastmilk or other liquid
  Interventions: Dietary Supplement: Thin liquid swallows
- Slightly thick liquid swallows (Experimental): Slightly thick liquid swallows of formula thickened with rice cereal or breastmilk or other liquid thickened with Gelmix
  Interventions: Dietary Supplement: Slightly thickened liquid swallows
- Mildly thick liquid swallows (Experimental): Mildly thick liquid swallows of formula thickened with rice cereal or breastmilk or other liquid thickened with Gelmix
  Interventions: Dietary Supplement: Mildly thickened liquid swallows
- Moderately thick liquid swallows (Experimental): Moderately thick liquid swallows of formula thickened with rice cereal or breastmilk or other liquid thickened with Gelmix
  Interventions: Dietary Supplement: Moderately thickened liquid swallows

INTERVENTIONS:
Dietary Supplement: Thin liquid swallows — Thin liquid swallows of formula or breastmilk or other liquid
  Arms: Thin liquid swallows
Dietary Supplement: Slightly thickened liquid swallows — Slightly thick liquid swallows of formula thickened with rice cereal or breastmilk or other liquid thickened with Gelmix
  Arms: Slightly thick liquid swallows
Dietary Supplement: Mildly thickened liquid swallows — Mildly thick liquid swallows of formula thickened with rice cereal or breastmilk or other liquid thickened with Gelmix
  Arms: Mildly thick liquid swallows
Dietary Supplement: Moderately thickened liquid swallows — Moderately thick liquid swallows of formula thickened with rice cereal or breastmilk or other liquid thickened with Gelmix
  Arms: Moderately thick liquid swallows

SUMMARY:
This study will examine the effects of varying liquid viscosity on swallow physiology in infants with oropharyngeal dysphagia and brief resolved unexplained event (BRUE) and other children with dysphagia that would be at risk for symptoms of swallow dysfunction.

DETAILED DESCRIPTION:
Infants with oropharyngeal dysphagia and in particular brief resolved unexplained events (BRUE) are a significant driver of pediatric health care expenditure since the mechanism for their swallow dysfunction is incompletely understood and therefore frequently goes unrecognized and untreated. We hypothesize that infants with oropharyngeal dysphagia and BRUE have measurable differences in swallowing physiology to explain their symptoms of cyanotic choking spells, that these differences can be quantified using pharyngeal high resolution impedance-manometry compared to videofluoroscopic swallow study results, and that this swallowing dysfunction can be safely corrected with a change of formula viscosity. Through this research project, we will systematically investigate the effects of thickened feedings on swallow function in infants with dysphagia and BRUE and perform detailed physiology studies on pharyngeal and esophageal motility as critical mediators of improved outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 0 to 21 years
* Admitted to Boston Children's Hospital after experiencing first lifetime BRUE, or with dysphagia symptoms such that they would be at risk for BRUE or other symptoms of swallowing difficulty
* Have had videofluoroscopic swallow study performed or might have future videofluoroscopic swallow study performed.

Exclusion Criteria:

* Any pre-existing medical diagnoses that exclude brief resolved unexplained event diagnosis including seizure disorders and cyanotic congenital heart disease
* Any nasal/pharyngeal/esophageal anomalies that might affect safe placement of the pharyngeal motility catheter
* Children fed exclusively by enteral tube
* Allergy to rice cereal or Gelmix thickener, which will be used to adjust liquid viscosity

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Swallow risk indices for thin vs mildly thick vs slightly thick liquids | 30 minutes
  We will calculate swallow risk index (SRI) from impedance-manometry results to compare mean SRI with thin liquids and thickened liquids for subjects with aspiration compared to mean SRI for thin liquids and thickened liquids in subjects without aspiration.

SECONDARY OUTCOMES:
Impedance-Manometry Swallow Physiology Metrics | 30 minutes
  We will measure swallow physiology metrics from impedance-manometry results, including post-swallow impedance ratio, to compare these parameters with thin liquids between subjects with and without aspiration and with varied liquid consistencies within subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Duncan, MD, MPH, Principal Investigator — Boston Children's Hospital; Rachel Rosen, MD, MPH, Study Director — Boston Children's Hospital; Sudarshan Jadcherla, MD, Study Director — Nationwide Children's Hospital; Taher Omari, PhD, Study Director — Flinders University; Samuel Nurko, MD, MPH, Study Director — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Duncan DR, Amirault J, Mitchell PD, Larson K, Rosen RL. Oropharyngeal Dysphagia Is Strongly Correlated With Apparent Life-Threatening Events. J Pediatr Gastroenterol Nutr. 2017 Aug;65(2):168-172. doi: 10.1097/MPG.0000000000001439. PMID 27741062
- [Background] Duncan DR, Larson K, Rosen RL. Clinical Aspects of Thickeners for Pediatric Gastroesophageal Reflux and Oropharyngeal Dysphagia. Curr Gastroenterol Rep. 2019 May 16;21(7):30. doi: 10.1007/s11894-019-0697-2. PMID 31098722
- [Background] Duncan DR, Growdon AS, Liu E, Larson K, Gonzalez M, Norris K, Rosen RL. The Impact of the American Academy of Pediatrics Brief Resolved Unexplained Event Guidelines on Gastrointestinal Testing and Prescribing Practices. J Pediatr. 2019 Aug;211:112-119.e4. doi: 10.1016/j.jpeds.2019.04.007. Epub 2019 May 15. PMID 31103259
- [Background] Rommel N, Selleslagh M, Hoffman I, Smet MH, Davidson G, Tack J, Omari TI. Objective assessment of swallow function in children with suspected aspiration using pharyngeal automated impedance manometry. J Pediatr Gastroenterol Nutr. 2014 Jun;58(6):789-94. doi: 10.1097/MPG.0000000000000337. PMID 24552674
- [Background] Omari TI, Dejaeger E, Van Beckevoort D, Goeleven A, De Cock P, Hoffman I, Smet MH, Davidson GP, Tack J, Rommel N. A novel method for the nonradiological assessment of ineffective swallowing. Am J Gastroenterol. 2011 Oct;106(10):1796-802. doi: 10.1038/ajg.2011.143. Epub 2011 May 10. PMID 21556039
- [Background] Duncan DR, Liu E, Growdon AS, Larson K, Rosen RL. A Prospective Study of Brief Resolved Unexplained Events: Risk Factors for Persistent Symptoms. Hosp Pediatr. 2022 Dec 1;12(12):1030-1043. doi: 10.1542/hpeds.2022-006550. PMID 36336644